CLINICAL TRIAL: NCT06119126
Title: Clinical Efficacy of SDF and Laser in Preventing Initial Caries Progression With and Without Fissure Sealants in Primary and Permanent Molars
Brief Title: Two Preventive Measures on Caries Progression in Mixed Dentition Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Islam el guindy, Assistant Lecturer in Pediatric Dentistry, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PED 20-3D
Record Dates: First submitted 2023-10-29; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Dentist's Role
Keywords: SDF; Diode Laser; Pits and fissure sealants; primary molars; permanent molars
MeSH Terms: interventions — silver diamine fluoride; Lasers, Semiconductor; Pit and Fissure Sealants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group A (Experimental): Diode laser application only
  Interventions: Device: Diode Laser
- Group B (Experimental): SDF application only
  Interventions: Drug: SDF1
- Group C (Experimental): Diode laser application followed by pits and fissure sealant.
  Interventions: Device: Diode Laser; Drug: Pit Fissure Sealant
- Group D (Experimental): SDF application followed by pits and fissure sealant.
  Interventions: Drug: SDF1; Drug: Pit Fissure Sealant

INTERVENTIONS:
Drug: SDF1 — Topical SDF application
  Other Names: silver diamine fluoride
  Arms: Group B; Group D
Device: Diode Laser — Irradiating Enamel by Diode laser
  Other Names: Class 4 dental laser
  Arms: Group A; Group C
Drug: Pit Fissure Sealant — Sealing occlusal pits and fissures
  Other Names: PFS
  Arms: Group C; Group D

SUMMARY:
Primary Objective:

Assessing the clinical effect of SDF and Laser on the prevention of initial caries progression with and without pits and fissure sealants in both permanent and primary molars.

Secondary Objective:

Effect of SDF and Laser Application on the subsequently applied pits and fissure sealants.

DETAILED DESCRIPTION:
Primary Objective:

Assessing the clinical effect of SDF and Laser on the prevention of initial caries progression with and without pits and fissure sealants in both permanent and primary molars.

Scoring caried out by ICDAS Scoring criteria over a 1 year follow up period

Secondary Objective:

Effect of SDF and Laser Application on the subsequently applied pits and fissure sealants.

Measured by Simonson's criteria over 1 year follow up period.

ELIGIBILITY:
Inclusion Criteria

.Children aged 6-9 years old.

.Patients categorized as moderate to high caries risk (deft index >1) showing more than 1 new carious lesions or restorations in the last 36 months according to "ADA Caries Risk Assessment Form (Age >6)" .A split mouth study design was followed where all four second molars were selected for intervention in the primary molar group, while all first molars were selected for intervention in the permanent molar group.

.The four molars selected in each patient (primary / permanent) should be fully erupted with no gingival overhangs /operculum and with no history of previous restorations or prior sealants.

.According to International Caries Detection and Assessment System ICDAS grading, molars with (0, 1, 2) scores only were included.

Exclusion Criteria:

.Uncooperative or mentally challenged patients, with bad oral hygiene or rampant caries.

.Patients providing history of bruxism or clenching affecting the posterior occlusion were excluded.

.Children with known allergies or sensitivities to resins or silver products. .Molars that showed well-coalesced, self-cleansing pits & fissures or shallow grooves and severe forms of hypoplasia / fluorosis were excluded.

.Patients & parents with high esthetic demands and concerns. .Unmotivated patients, or parents who refused to sign the consent form.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Number of molars with arrested initial decay | 1 year follow up
  ICDAS II Score system

SECONDARY OUTCOMES:
Number of molars with completely retained f pits and fissure sealants | 1 year follow up
  Simonsen's Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Noha Kabil, Professor, Study Director — Head of Department; Basma Gamal, Lecturer, Study Director — Faculty Council Member
Locations (1):
- Faculty of Dentistry British University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No